CLINICAL TRIAL: NCT00132262
Title: Brief Intervention to Reduce Injury in Minorities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Raul Caetano, Professor - School of Public Health, Dallas Regional Campus, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: R01AA013824 (NIH)
Record Dates: First submitted 2005-08-16; First posted 2005-08-19 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Injuries; Alcohol Related Disorders
Keywords: Screening and Brief Intervention; Ethnic Differences; Trauma Center
MeSH Terms: conditions — Wounds and Injuries; Alcohol-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients randomized to this arm received an intervention based in the motivational interviewing style
  Interventions: Behavioral: Brief intervention based on motivational interviewing
- 2 (Active Comparator): Patients randomized to this arm received standard hospital care
  Interventions: Behavioral: Standard Care including referral for treatment

INTERVENTIONS:
Behavioral: Brief intervention based on motivational interviewing — The intervention was an approximately 30 minute discussion about alcohol-related risk behaviors and motivation to change
  Arms: 1
Behavioral: Standard Care including referral for treatment — Standard hospital care provided the patient with information and referral for treatment as necessary.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effectiveness and ethnic differences of a brief alcohol intervention for injured patients.

DETAILED DESCRIPTION:
Injuries are not isolated events or one time occurrences and injury has been identified as an important public health problem. Among the risk factors associated with injury and injury recidivism, the most widely recognized is alcohol use with approximately 50% of all injuries associated with alcohol. In general, alcohol use and drinking patterns vary by ethnicity, with frequent heavy drinking and associated problems more common among Blacks and Hispanics. Blacks, in general, suffer a disproportionate level of alcohol problems, despite having higher rates of abstention than Whites and Hispanics. Hispanics also generally suffer more alcohol-related problems than whites. Overall, injury recidivism is higher among poorer, minority populations and among individuals who abuse alcohol. The efficacy of brief alcohol interventions in the emergency care setting such as hospital emergency departments and trauma care centers is a relatively new area of research. Brief alcohol interventions appear to reduce alcohol intake and rates of injury following hospitalization; however, there is a need to evaluate the efficacy of these brief interventions in various ethnic groups. The proposed research involves a randomized controlled trial of a brief alcohol intervention based upon motivational interviewing and harm reduction to reduce alcohol consumption and injury following admission to an emergency room or trauma department for treatment of an injury. The primary aim of the proposed project is to determine the efficacy of this intervention as applied in the trauma care and emergency room setting among Whites, Blacks and Hispanics. The three outcomes of interest include:

1. alcohol consumption as measured by number of standard drinks consumed per week and
2. frequency of drinking five or more drinks per occasion engagement in injury related risk behaviors and
3. injury recidivism rates

It is hypothesized that the brief alcohol intervention will have a greater impact on alcohol consumption, injury related risk behaviors and injury recidivism among Whites than Blacks and Mexican Americans. In addition, it is hypothesized that the brief alcohol intervention will have less of an impact on alcohol consumption, injury related risk behaviors and injury recidivism among Mexican Americans born in the United States than among those born in Mexico after controlling for acculturation, acculturation stress and sociodemographic characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Admission for treatment of an injury
* Self identification of Black, White or Hispanic Ethnicity
* Age > 17
* Screen positive for potential alcohol related injury based upon clinical indication of alcohol use prior to injury including positive blood alcohol concentration, self report of alcohol use prior to injury, heavy drinking or drinking beyond normal limits as defined by NIAAA

Exclusion Criteria:

* Glasgow Coma Score or GCS < 14
* Admission for self inflicted injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1493 (Actual)
Dates: Start 2003-05; Primary Completion 2006-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
alcohol intake | six months and one year
injury recidivism | six months and one year

SECONDARY OUTCOMES:
alcohol problems | six months and one year
injury related risk behaviors | 6 months and one year

CONTACTS AND LOCATIONS:
Overall Officials: Raul Caetano, MD, PhD, Principal Investigator — University of Texas Health Science Center School of Public Health Dallas Campus

REFERENCES:
- [Derived] Cochran G, Field C, Caetano R. Injury-related consequences of alcohol misuse among injured patients who received screening and brief intervention for alcohol: a latent class analysis. Subst Abus. 2014;35(2):153-62. doi: 10.1080/08897077.2013.820679. PMID 24821352
- [Derived] Cochran G, Field C, Caetano R. Changes in Classes of Injury-Related Risks and Consequences of Risk-Level Drinking: a Latent Transition Analysis. J Behav Health Serv Res. 2015 Jul;42(3):355-66. doi: 10.1007/s11414-013-9378-3. PMID 24259197
- [Derived] Field CA, Caetano R, Harris TR, Frankowski R, Roudsari B. Ethnic differences in drinking outcomes following a brief alcohol intervention in the trauma care setting. Addiction. 2010 Jan;105(1):62-73. doi: 10.1111/j.1360-0443.2009.02737.x. Epub 2009 Nov 17. PMID 19919597